CLINICAL TRIAL: NCT04190706
Title: Synergistic Innovative Functional Food Concepts to Neutralize Inflammation for Cardiometabolic Risk Prevention.
Acronym: SINFONI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 69HCL18_0097
Record Dates: First submitted 2019-11-13; First posted 2019-12-09 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Cardiometabolic Risk; Abdominal Obesity
Keywords: inflammation; cardiometabolic risk; endotoxemia; polyphenols; oxidative stress; slow digestible starch; fibers; gut microbiota; nutritional challenge test
MeSH Terms: conditions — Obesity, Abdominal; Inflammation; Endotoxemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- bioactive components fortified food products (Experimental)
  Interventions: Other: bioactive components fortified food products intake (biscuits and cookies)
- control food products (Placebo Comparator)
  Interventions: Other: control food products intake (biscuits and cookies)

INTERVENTIONS:
Other: bioactive components fortified food products intake (biscuits and cookies) — Volunteers will have to consume daily 100 g of fortified biscuits and cookies instead of those usually consumed during nine weeks. The last week, volunteers will have to consume daily a fructose solution (3g/kg fat free mass)
  Arms: bioactive components fortified food products
Other: control food products intake (biscuits and cookies) — Volunteers will have to consume daily 100 g of standard biscuits and cookies instead of those usually consumed during nine weeks. The last week, volunteers will have to consume daily a fructose solution (3g/kg fat free mass)
  Arms: control food products

SUMMARY:
The aim of the study is to evaluate the synergistic effects of daily consumption of food products fortified with bioactive components (fibres, polyphenols, omega-3, Slow Digestible Starch) for 9 weeks, compared to the daily intake of standard food products on low-grade inflammation in cardiometabolic risk subject.

The inflammatory parameters will be assessed in fasting and in postprandial period after the consumption of a hyper-carbohydrate and hyper-lipidic test meal called Flexmeal. A metabolic stress will be induced by a fructose ingestion challenge during the last 6 days of interventional period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Body Mass Index of 25 to 35 kg/m2
* Waist circumference greater than 80 cm for women and than 96 cm for men
* Daily biscuits consumption
* Fibers intake <25g/day

Exclusion Criteria:

* Medical history of digestive surgery or disease
* Large polyphenols food products consumer (cranberries, red berries, coffee, tea, red wine, fruits and vegetables…)
* Current or recent (<12 weeks) intake of antibiotics or gastro-intestinal medicinal product
* Current probiotics, prebiotics, fibers complement, and/or any products modulation gut transit
* Feeding particular diet such as vegetarian diet or hyperprotein diet
* Current weight loss diet
* Pregnant or lactating woman or woman who did not use effective contraception
* Drinking more than 3 glasses of alcohol per day (>30g/day)
* Smoking more than 5 cigarettes per day

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Change from baseline postprandial plasma endotoxemia binding protein kinetics: LBP (lipopolysaccharide-binding protein) and CD14 (Cluster of differentiation 14) | baseline, 8 and 9 weeks
  LBP and CD14 proteins will be measured at time 0, 120 and 300 after test meal intake

SECONDARY OUTCOMES:
Change from baseline fasting and postprandial plasma inflammatory markers: MCP-1, RANTES, IFNγ, IL-6, TNF-α, IL-1β, CRPus, adiponectin | baseline, 8 and 9 weeks
  MCP-1 ( monocyte chemotactic protein-1), RANTES (Regulated on activation, normal T expressed and secreted), IFNγ (Interferon γ) , IL-6 (Interleukin 6), TNF-α (Tumor Necrosis Factor α), IL-1β (Interleukin 1β), CRPus, adiponectin will be measured at time 0 and 300 minutes after test meal intake
Change of fasting and postprandial plasma inflammatory endotoxemia LPS (lipopolysaccharide) | baseline, 8 and 9 weeks
  LPS will be measured at time 0, 60, 120, 180, 240, 300 after test meal intake
Change from baseline fasting and postprandial plasma endothelial function markers: Human CVD Panel 2, Lipocalin-2/NGAL, Myeloperoxidase, sICAM-1, sVCAM-1, ADAMTS13, D-dimer, GDF-15, Myoglobin, sP-Selectin, Serum Amyloid A | baseline, 8 and 9 weeks
  Human CVD Panel 2, Lipocalin-2/NGAL (neutrophil gelatinase-associated lipocalin), Myeloperoxidase, sICAM-1(Soluble Inter-cellular Adhesion Molecule-1), sVCAM-1(Soluble Form of Vascular Cell Adhesion Molecule 1), ADAMTS13 (a disintegrin and metalloproteinase with a thrombospondin type 1 motif, member 13), D-dimer, GDF-15 (Growth differentiation factor 15), Myoglobin, sP-Selectin, Serum Amyloid A will be measured at time 0 and 300 minutes after test meal intake
Change from baseline fasting plasma oxidative stress parameters: GSH, GSSG, Glutathion peroxidase/ reductase activity, MDA | baseline, 8 and 9 weeks
  GSH (glutathione), GSSG (glutathione disulfide), Glutathion peroxidase/ reductase activity will be measured at time 0 and MDA (malondialdehyde) will be measured at 0 and 300 minutes after test meal intake
Change from baseline body composition | baseline, 8 and 9 weeks
  Body composition will be measured by BodPod technique
Change from baseline plasma metabolites and hormone kinetics : glucose, insulin, triglycerides, non-esterified fatty acids | baseline, 8 and 9 weeks
  Plasma metabolites and hormone will be measured at time -30, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 minutes after test meal intake
Change from baseline fasting plasma lipids : total cholesterol , HDL cholesterol, LDL cholesterol, triglycerides, non-esterified fatty acids | baseline, 8 and 9 weeks
  fasting plasma lipids will be measured before test meal ingestion
Change from baseline resting energy expenditure | baseline, 8 and 9 weeks
  resting metabolic rate will be measured by indirect calorimetry
Change from baseline substrates oxidation | baseline, 8 and 9 weeks
  substrates oxidation will be measured by indirect calorimetry after test meal intake during five hours.
Change from baseline gut microbiota composition | baseline, 8 weeks
  gut microbiota composition will be measured by 16S RNA (ribonucleic acid) analysis
Change from baseline stool consistency | nine weeks
  stool consistency will be measured by Bristol scale and every week during the interventional period
Change from baseline stool frequency | nine weeks
  stool frequency will be measured by questionnaire at baseline and every week during the interventional period
Change from baseline tolerance gastro-intestinal symptoms like bloating ,abdominal rumbling ,flatulence ,abdominal pain, nausea, vomiting | nine weeks
  Gastro intestinal symptoms will be collected by questionnaires and visual analogue scale (VAS) score (on a 90mm horizontal line; from no symptom (minimal) to serious symptom (maximum)) at baseline and every week during the interventional period
Change from baseline diet intake | baseline, 8 and 9 weeks
  diet intake will be evaluated by a three days diet survey
Change from baseline fasting plasma zonulin | baseline, 8 and 9 weeks
  comparison of fasting plasma zonulin from baseline
Change from baseline polyphenols urinary concentrations | baseline, 8 weeks
  Comparison of polyphenols urinary concentrations from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Martine LAVILLE, Pr, Principal Investigator — Centre de Recherche en Nutrition Humaine Rhône-Alpes
Locations (1):
- Centre de Recherche en Nutrition Humaine Rhône-Alpes, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hornero-Ramirez H, Morisette A, Marcotte B, Penhoat A, Lecomte B, Panthu B, Lessard Lord J, Thirion F, Van-Den-Berghe L, Blond E, Simon C, Caussy C, Feugier N, Dore J, Sanoner P, Meynier A, Desjardins Y, Pilon G, Marette A, Cani PD, Laville M, Vinoy S, Michalski MC, Nazare JA. Multifunctional dietary approach reduces intestinal inflammation in relation with changes in gut microbiota composition in subjects at cardiometabolic risk: the SINFONI project. Gut Microbes. 2025 Dec;17(1):2438823. doi: 10.1080/19490976.2024.2438823. Epub 2024 Dec 22. PMID 39710576
- [Background] Demangeat A, Hornero-Ramirez H, Meynier A, Sanoner P, Atkinson FS, Nazare JA, Vinoy S. Complementary Nutritional Improvements of Cereal-Based Products to Reduce Postprandial Glycemic Response. Nutrients. 2023 Oct 17;15(20):4401. doi: 10.3390/nu15204401. PMID 37892479